CLINICAL TRIAL: NCT00819845
Title: Effects of Cardioprotective Therapy, Carvedilol vs Ramipril, in Patients Affected by Duchenne and Becker Muscular Dystrophy. Clinical Significance and Prognostic Value of Cardiac Magnetic Resonance Study.
Brief Title: Ramipril Versus Carvedilol in Duchenne and Becker Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Catholic University, Italy (Other)
Responsible Party: Vincenzo Giglio MD, PhD, Uildm of Rome
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Uildm Rome
Record Dates: First submitted 2009-01-08; First posted 2009-01-09 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2009-01

CONDITIONS: Duchenne Muscular Dystrophy; Becker Muscular Dystrophy
Keywords: Duchenne; Becker muscular dystrophy; cardioprotective therapy; cardiac magnetic resonance; ultrasound tissue characterization
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — Carvedilol; Adrenergic beta-Antagonists; Ramipril; Angiotensin-Converting Enzyme Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ramipril (Experimental)
  Interventions: Drug: ramipril
- Carvedilol (Experimental)
  Interventions: Drug: carvedilol

INTERVENTIONS:
Drug: carvedilol — carvedilol vs ramipril
  Other Names: Beta-Blocker
  Arms: Carvedilol
Drug: ramipril — carvedilol vs ramipril
  Other Names: ACE-inhibitor
  Arms: Ramipril

SUMMARY:
Data on preventive therapy in Duchenne muscular dystrophy (DMD) and Becker muscular dystrophy (BMD) affected individuals without cardiac involvement are very limited and currently lacking regard both ACE-inhibitors and Beta-Blockers in Becker Muscular Dystrophy and for the latter even in Duchenne Muscular Dystrophy patients. Thus, the study aim is to compare the efficacy of carvedilol vs ramipril on myocardial tissue properties and heart function, performing CMR and myocardial Ultrasound Tissue Characterisation analysis.

DETAILED DESCRIPTION:
This protocol represent an open randomized and prospective trial, designed to answer the specific question regarding the role of the cardioprotective therapy in Duchenne Muscular Dystrophy and Becker Muscular Dystrophy patients. In this light, CMR could provide relevant data, reinforcing the scientific background, to start early (particularly in BMD patients in whom this is still a debated question) a cardioprotective treatment with carvedilol or ramipril.Finally,this clinical trial will clarify whether a preventive therapy may be helpful on the clinical outcome, both in reducing myocardial fibrosis and preventing the progression towards the cardiomyopathy.

ELIGIBILITY:
Inclusion Criteria:

1. Immunohystochemical and molecular diagnosis of Duchenne and Becker muscular dystrophy.
2. Not evidence of clinical cardiomyopathy,normal 2D-echocardiography with normal systolic,WMSI = 1) and diastolic function.
3. DMD patients treated with steroid therapy.
4. All DMD and BMD patients are not treated with cardiological therapy (ACE-inhibitors, ARBs or Beta-Blockers).
5. Written informed consent to study participation (with serial visit, CMR and echocardiographic study) is required from all patients themselves, as well as their parent or guardian and healthy-control subjects.

Exclusion Criteria:

1. Failure to obtain informed consent from patients, parents or guardians.
2. Any controindications to carvedilol or ramipril treatment (bronchial asthma, diabetes, any degree of renal failure (all patients are required to have a normal creatinine level and clearance).
3. in BMD patients ECG changes suggestive of ischemic heart disease, left bundle-branch block, atrial flutter/fibrillation, ventricular arrhythmias, any degree of atrioventricular block and left ventricular (LV) hypertrophy. Aspecific ST changes will be not considered as electrocardiographic exclusion criteria both in DMD and BMD patients.
4. In BMD patients exclusion criteria will be also hypertension and valvular heart disease other than trivial.
5. DMD and BMD patients requiring ventilatory (non-invasive or invasive) assistance.
6. Presence of systolic and/or diastolic dysfunction detected by 2D-Echocardiography.
7. Presence of any contraindications to CMR (including any history of claustrophobia).
8. Patients under the age of 2 years.
9. Renal failure, even mild.
10. Patient unable or unwilling to attend the follow-up and tests, in the opinion of local study principal investigator, (children not willing to perform CMR will not be enrolled).

Ages: 2 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 194 (Estimated)
Dates: Start 2008-12; Primary Completion 2009-06 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Left ventricular Ejection Fraction, systolic and diastolic left ventricular volumes and LGE (as a quantitative measure) detected by MRI and myocardial Ultrasound Tissue Characterisation data by Echocardiography. | 1 year

SECONDARY OUTCOMES:
Prevalence of LGE in DMD and BMD patients,the effects of pharmacological therapy both on LGE evolution and myocardial UTC analysis. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Giglio, MD, PhD, Principal Investigator — Uildm, Rome
Locations (1):
- Unione Italiana lotta Distrofia Muscolare, Rome, Italy